CLINICAL TRIAL: NCT06801769
Title: Study for the Identification of a Quantitative Eco-Elastographic Score of Pancreatic Steatosis and Its Correlation with Beta-Cell Function and Metabolic Syndrome.
Brief Title: Study for the Identification of a Score to Assess Intrapancreatic Fat Through Eco-Elastography and Its Correlation with Metabolic Syndrome and Insulin-Secreting Cells.
Acronym: SPES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Teresa Mezza, M.D, PhD, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 7291
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Pancreatic Steatosis; Metabolic Syndrome X; Diabetes Mellitus
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients Undergoing Endoscopic Ultrasound (Experimental)
  Interventions: Diagnostic Test: C-peptide

INTERVENTIONS:
Diagnostic Test: C-peptide — Measurement of C-peptide at 5 time points during a standard oral glucose tolerance test (OGTT).

SUMMARY:
**Brief Summary of the SPES Clinical Study**

The SPES clinical study aims to evaluate the relationship between pancreatic fat accumulation (pancreatic steatosis) and metabolic health. Pancreatic steatosis has been linked to conditions like type 2 diabetes (T2D) and metabolic syndrome, but the underlying mechanisms and its impact on beta-cell function remain poorly understood.

The primary goal of this study is to develop a quantitative ultrasound elastography score to measure the degree of pancreatic steatosis and explore how this relates to pancreatic beta-cell function and key factors associated with the development of type 2 diabetes and metabolic syndrome.

A secondary goal is to categorize participants into four risk classes for type 2 diabetes based on their metabolic profiles and correlate these classes with the degree of pancreatic steatosis. This may provide insights into individual risk stratification for T2D and related complications.

The study will enroll 100 participants, aged 18 to 80, attending the Endoscopic Ultrasound Unit at the Fondazione Policlinico Universitario Agostino Gemelli in Rome. Participants will undergo endoscopic ultrasound for various clinical reasons, excluding those with pancreatic tumors, cystic fibrosis, or insulin-treated diabetes. Key inclusion criteria include controlled blood glucose levels (HbA1c < 10% or fasting glucose < 250 mg/dL) and the ability to understand and provide informed consent.

The study is interventional but does not involve drugs or medical devices. Participants will attend a visit where medical history, physical measurements (e.g., BMI, waist circumference, blood pressure), glucose tolerance tests, and blood work will be collected. This comprehensive approach aims to better understand the metabolic implications of pancreatic steatosis and its role in type 2 diabetes development.

The study will last 24 months, including the enrollment period. Findings may contribute to improved risk stratification, prevention, and management strategies for type 2 diabetes and related conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* HbA1c <10% or fasting glucose <250 mg/dL
* Ability to understand and provide informed consent regarding the procedures, data collection, and analysis.

Exclusion Criteria:

* Age <18 years or >80 years
* History of diabetes treated with insulin
* HbA1c >10% or fasting glucose >250 mg/dL
* Pancreatic diseases (solid tumors/secretory NETs/cystic fibrosis; non-secretory NETs and IPMN may be included)
* Previous pancreatic surgery
* Moderate anemia (Hb <10 mg/dL)
* Severe liver failure (Child-Pugh C)
* Non-metabolic causes of NAPLD (e.g., corticosteroid therapy, antiretrovirals, gemcitabine, octreotide, history of hemochromatosis, malnutrition, HBV/HIV infections)
* Alcohol abuse (>30 g/day of ethanol)
* Pregnancy and breastfeeding
* Inability to adequately understand informed consent and study procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Identification of a quantitative ultrasound elastography score for the degree of pancreatic steatosis | One day assessment

SECONDARY OUTCOMES:
Correlation of the score with metabolic and functional parameters across the four different risk classes for type 2 diabetes. | One day assessment